CLINICAL TRIAL: NCT05306600
Title: Onco-Genomas Brasil: Mapping Breast and Prostate Cancer in the Brazilian Public Health System
Status: Recruiting | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: 55457122.3.0000.5330
Record Dates: First submitted 2022-03-09; First posted 2022-04-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: breast cancer; prostate cancer; exome
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and formalin-fixed paraffin-embedded (FFPE) tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer: 745 patients with HER2-positive and triple-negative breast cancer who underwent neoadjuvant therapy followed by breast surgery.
  Interventions: Diagnostic Test: whole exome and whole genome sequencing analysis
- Prostate cancer: 137 patients with metastatic prostate cancer
  Interventions: Diagnostic Test: whole exome and whole genome sequencing analysis

INTERVENTIONS:
Diagnostic Test: whole exome and whole genome sequencing analysis — Somatic and germline whole exome sequencing will be analyzed for prostate and HER2-positive breast cancer
  Somatic whole exome and germline whole genome sequencing will be analyzed for triple-negative breast cancer

SUMMARY:
This project aims to perform complete sequencing of the somatic (tumor) and germline exomes during clinical investigation of cancer patients treated through the Brazilian Unified Health System to generate genomic and phenotypic data for the Brazilian Ministry of Health's National Precision Genomics and Health Program, called Genomas Brasil, as well as to collect data on the population's ancestry.

DETAILED DESCRIPTION:
In Brazil, the most frequent types of neoplasm are prostate cancer in men and breast cancer in women. Understanding the molecular variants in tumors, which result from mutations and variants that occur during carcinogenesis, can affect treatment response and disease prognosis and is an important target of oncology research. Detecting hereditary genetic syndromes also helps in oncological follow-up, allowing prediction of the risk of new neoplasms. This project aims to perform complete sequencing of the somatic (tumor) and germline exomes during clinical investigation of cancer patients treated through the Brazilian Unified Health System to generate genomic and phenotypic data for the Brazilian Ministry of Health's National Precision Genomics and Health Program, called Genomas Brasil, as well as to collect data on the population's ancestry.

ELIGIBILITY:
Inclusion criteria for breast cancer patients (Arm 1):

* Women aged ≥ 18 years;
* Brazilian nationality;
* After review at the Hospital Moinhos de Vento, confirmed histological diagnosis of breast carcinoma with overexpression of HER2 (classified by immunohistochemistry as 3+ or 2+ with positive in-situ hybridization) or triple-negative (estrogen and progesterone receptors <1% and no overexpression of HER2);
* Clinical stage II or III for HER2-positive and I, II and III for triple-negative patients - American Joint Committee on Cancer (AJCC) 8th edition;
* HER2- positive patients: must undergo neoadjuvant chemotherapy plus trastuzumab in the following regimens: anthracycline (doxorubicin or epirubicin) followed by taxane (docetaxel or paclitaxel), combined with trastuzumab, or a non-anthracycline option consisting of taxane (docetaxel or paclitaxel) combined with carboplatin and trastuzumab;
* Triple-negative patients: must undergo neoadjuvant chemotherapy without immunotherapy in the following regimens: anthracycline (doxorubicin or epirubicin) followed by taxane (docetaxel or paclitaxel) with/ without platins (carboplatin ou cisplatin) or a regimen without anthracycline (taxane with/without platins)
* Patients must provide written informed consent prior to inclusion

Inclusion criteria for patients with prostate cancer (Arm 2):

* Men aged ≥ 18 years;
* Confirmed histological diagnosis of prostate adenocarcinoma;
* AJCC 8th edition clinical stage IV;
* Patients must provide written informed consent.

Exclusion criteria for Arms 1 and 2:

* No available paraffin-embedded tumor tissue for genomic analysis;
* Inability to collect blood for genomic evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Institutions from each region that serve Public Health System patients and have high complexity oncology care centers will be included in both Arms to provide a sample that represents the heterogeneity of the Brazilian population. Institutions previously evaluated and validated by the Brazilian Ministry of Health will be selected after completing a feasibility questionnaire. It is estimated that 25 to 30 institutions will be included (at least one from each region) in Arm 1. For Arm 2, 10 centers will be selected from among previously approved institutions.
Sampling Method: Non-Probability Sample
Enrollment: 882 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize complete somatic and germline exomes/genomes in a Brazilian population | 12 months
  Mutations in the somatic and germline exomes/genomes of women with HER2-positive and triple-negative breast cancer and of men with metastatic prostate cancer will be described

SECONDARY OUTCOMES:
To identify genetic variants related to tumor prognosis | 12 months
  Mutations in the somatic and germline exomes/genomes will be correlated to clinical outcomes
To identify genetic variants predictive of response to treatments | 12 months
  Mutations in the somatic and germline exomes/genomes will be correlated to response to treatments
Number of patients with mutations in cancer-predisposing genes | 12 months
  Identify mutations in germline exomes/genomes related to hereditary cancer syndromes

OTHER OUTCOMES:
To identify the ancestry of patients with breast and prostate cancer | 12 months
  Characterize the genomic ancestry of Brazilian patients with breast and prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Daniela D Rosa, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (19):
- Brazil (19):
  - Hospital Universitário Getúlio Vargas, Manaus, Amazonas
  - Hospital Santa Rita de Cássia - AFECC, Vitória, Espírito Santo
  - Hospital Calixto Midlej Filho/ Santa Casa de Itabuna, Itabuna, Estado de Bahia
  - Hospital do Câncer do Maranhão, São Luís, Maranhão
  - Hospital da Santa Casa de Misericórdia, Belo Horizonte, Minas Gerais
  - Hospital das Clínicas, Belo Horizonte, Minas Gerais
  - Hospital do Câncer/União Oeste Paranaense de Estudo e Combate ao Câncer, Cascavel, Paraná
  - Hospital Universitário João de Barros Barreto, Belém, Pará
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital Escola da Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - Hospital do Amor, Barretos, São Paulo
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Hospital Araújo Jorge, Goiânia
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Grupo Hospitalar Conceição, Porto Alegre
  - Hospital Fêmina, Porto Alegre
  - Hospital São Camilo, São Paulo
  - Hospital Universitário Cassiano Antônio de Moraes, Vitória

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schuch JB, Bordignon C, Rosa ML, de Baumont AC, Bessel M, Macedo GS, Rosa DD. Mapping breast and prostate cancer in the Brazilian public health system: study protocol of the Onco-Genomas Brasil. Front Oncol. 2024 Mar 13;14:1350162. doi: 10.3389/fonc.2024.1350162. eCollection 2024. PMID 38544834